CLINICAL TRIAL: NCT02023229
Title: High-fiber High-fiber Diet and Branched Chain Aminoacids. Impact on Nutritional Status and Complications in Patients With Liver Cirrhosis
Brief Title: Branched Chain Aminoacid Supplementation in Patients With Liver Cirrhosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, ALDO TORRE DELGADILLO, Principal investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Enterex01
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Liver Cirrhosis
Keywords: Branched chain aminoacids; Nutritional status; Hepatic encephalopathy
MeSH Terms: conditions — Liver Cirrhosis; Hepatic Encephalopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diet plus branched chain aminoacids (Experimental): High-fiber high-protein diet Oral supplement : branched chain aminoacids
  Interventions: Dietary Supplement: Branched-chain aminoacids; Other: High-fiber high protein diet
- Diet (Active Comparator): High-fiber high-protein diet
  Interventions: Other: High-fiber high protein diet

INTERVENTIONS:
Dietary Supplement: Branched-chain aminoacids
  Arms: Diet plus branched chain aminoacids
Other: High-fiber high protein diet

SUMMARY:
Malnutrition is a frequent complication in patients with liver cirrhosis. Most patients have decreased dietary intake due to ascites, hepatic encephalopathy and pro-inflammatory cytokines.

We hypothesized that branched chain aminoacids can improve nutritional status and delay episodes of hepatic encephalopathy

ELIGIBILITY:
Inclusion Criteria:

Ambulatory patients Patients with confirmed diagnose of liver cirrhosis Patients classified as Child-Pugh A or Child Pugh B

Exclusion Criteria:

Acute or chronic renal failure Pregnancy Overt hepatic encephalopathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Nutritional status | At time of recruitment
  Assessed by bioelectrical impedance vector analysis and mid-arm muscle circumference

SECONDARY OUTCOMES:
Hepatic Encephalopathy | At time of recruitment

OTHER OUTCOMES:
Nutritional status | 3 months follow-up
  Assessed by bioelectrical impedance vector analysis and mid-arm muscle circumference
Nutritional status | 6 months follow-up
  Assessed by bioelectrical impedance vector analysis and mid-arm muscle circumference
Hepatic encephalopathy | 6 months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición "Salvador Zubirán", Mexico City, Mexico